CLINICAL TRIAL: NCT00660452
Title: A Randomised, Double-blind, Placebo-controlled, Multi-centre, Phase III Study to Assess Efficacy and Safety of STALORAL® 300 IR Sublingual Immunotherapy (SLIT) in Chinese Asthmatic Patients Allergic to House-dust Mites
Brief Title: A Phase III Study to Assess Efficacy and Safety of STALORAL® 300 IR Sublingual Immunotherapy (SLIT) in Asthmatic Patients Allergic to House-dust Mites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VO55.06 CHIN
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Allergy
Keywords: Allergy; SLIT; Asthma; House Dust Mites
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 360 active patients with house dust mites related asthma with or without allergic rhinitis
  Interventions: Drug: Staloral
- 2 (Placebo Comparator): 180 patients in the placebo group with house -dust mites related asthma with or without allergic rhinitis.
  Interventions: Drug: Staloral

INTERVENTIONS:
Drug: Staloral — Sublingual immunotherapy with Staloral dust mites solution

SUMMARY:
A phase III study to assess the efficacy and safety of sublingual immunotherapy with STALORAL dust mites solution compared with placebo for reduction of asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients aged 16 to 50 years (inclusive).
2. House dust mite-induced allergic asthma with or without perennial allergic rhinitis for at least 1 year.
3. Sensitised to D. pteronyssinus and D.farinae (positive skin prick test (SPT) with wheal diameter ≥ 4 mm and specific IgE level ≥ 0.70 kU/L
4. Patients treated with inhaled corticosteroids (ICS) before the screening visit at a dose ≥ 200 µg and < 1,000 µg equivalent budesonide/day.

Exclusion Criteria:

1. Mild intermittent asthma needed to be treated only with β2-agonist (GINA level 1).
2. Severe asthma needed to be treated with inhaled corticosteroids with a dose ≥ 1,000 µg/day equivalent budesonide.
3. FEV1 < 70% of predicted value at Visit 1.
4. Co-sensitisation to other inhalant allergens than dust mites leading to clinically relevant allergic asthma and proven by a positive skin prick test with wheal diameter ≥ 4 mm and serum specific IgE ≥ 0.70 KU/L .
5. Patients with a past or current disease, which as judged by the investigator, may affect the patient's participation in or the outcome of the study. These diseases include, but are not limited to, past or current cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, immunological disease and endocrine disease.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 484 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
determine the proportion of patients who achieve well-controlled asthma with SLIT compared to placebo | September 2009

SECONDARY OUTCOMES:
Daily dose of steroids at the endpoint Number of asthma exacerbations Asthma Control Questionnaire(ACQ)score Asthma Quality of Life Questionnaire (AQLQ) score Lung Function Parameters ( FEV1; FEF 25-75 %; PEF) Allergic rhinitis g | September 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jia YIN, Pr., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital -, Beijing, China

REFERENCES:
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419
- [Derived] Devillier P, Fadel R, de Beaumont O. House dust mite sublingual immunotherapy is safe in patients with mild-to-moderate, persistent asthma: a clinical trial. Allergy. 2016 Feb;71(2):249-57. doi: 10.1111/all.12791. Epub 2015 Nov 6. PMID 26465232
- [Derived] Wang L, Yin J, Fadel R, Montagut A, de Beaumont O, Devillier P. House dust mite sublingual immunotherapy is safe and appears to be effective in moderate, persistent asthma. Allergy. 2014 Sep;69(9):1181-8. doi: 10.1111/all.12188. Epub 2014 Jul 24. PMID 25056584